CLINICAL TRIAL: NCT03671317
Title: Effect of Medical Clown Intervention on Anxiety and Perceived Pain Levels in Pediatric Patients Undergoing Venous Blood Draw
Brief Title: Medical Clowns for Pediatric Blood Draw
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Brent Blair, PhD, Director, Institute for Theatre & Social Change, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APP-18-03557
Record Dates: First submitted 2018-08-27; First posted 2018-09-14 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Anxiety State; Pain; Stress
Keywords: palliative care; medical clowning; anxiety relief; pain reduction; distraction; humor; papoose; restraints
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Participants are randomized to either receive medical clowning intervention or no intervention. The total length of subject participation is the participant's one visit to the blood draw clinic. Data collection involves pre then post surveys to measure anxiety and pain levels for comparison.
  After screening, consent, and randomization, the participants and legal guardians assigned to both arms will complete a survey. Once completed, the intervention arm is introduced to two medical clowns who accompany the participant through the blood draw process. The non intervention arm will continue with usual care. Audio recording begins when participants of both arms enter the blood draw room. Once the nurse leaves the room after venipuncture, all participants and legal guardians complete a second questionnaire.
  At the conclusion of the study, the medical staff are asked to answer a questionnaire rated on the Likert Scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This arm will receive a medical clowning intervention in addition to pre and post surveys about the blood draw process.
  Interventions: Behavioral: Medical Clowning
- Non-intervention group (No Intervention): This arm will continue usual care with no intervention from medical clowns. They will be asked to complete pre and post surveys about the blood draw process.

INTERVENTIONS:
Behavioral: Medical Clowning — This arm will receive a medical clowning intervention in addition to pre and post surveys about the blood draw process.
  Arms: Intervention group

SUMMARY:
The research objective of this proposed clinical trial is to determine the efficacy of a medical clowning intervention for pediatric patients undergoing venipuncture. Efficacy is defined in terms of decreasing anxiety, pain, and crying duration, and increasing the pace and ease of the procedure. The study population includes pediatric patients between the ages of 3 - 11 years who must undergo venipuncture at the LAC + USC Outpatient Clinic. The subjects will be randomized into two groups. The control subjects will receive no intervention during blood draw, while the intervention subjects will receive the medical clown intervention during blood draw. The clowns will interact with one patient at a time, engaging in play with the patient and caretakers during all parts of the procedure. Duration of crying and the duration of the entire procedure, the patient's level of pain and anxiety, the caretaker's level of anxiety, need for restraining devices (papoose) and the efficiency of the procedure will be measured. In order to perform the survey and self-assessment procedures, we will implement the use of measurement scales including a novel "emoji" child distress assessment scale, and a published adult anxiety scale (State-Trait Anxiety Inventory Form Y-1). The data will be analyzed using descriptive statistics.

DETAILED DESCRIPTION:
The scientific aim of this project is to determine the effect a medical clowning intervention may have on perceived pain levels and anxiety levels with patients, their families, and the medical staff during routine blood draw procedures in the Pediatric Oncology Hematology Clinic of LAC + USC.

We are investigating the following claims: First, the physical, play-based, non-verbal based forms of communication that a clown implements is effective in creating playful distraction during the procedure. The presence of the clown in this capacity can meaningfully reduce perceived pain levels in patients during venipuncture and reduce the duration of crying. Second, the clown intervention decreases anxiety levels in the trial participants and families leading up to and during blood draw which supports the patient as well as increases efficiency for hospital staff. Third, the presence of the clown will significantly reduce physical restraint (i.e. medical stabilization board, known as a papoose board) usage during venipuncture. Lastly, we aim to prove that coulrophobia does not play a factor in medical clowning interventions.

The USC School of Dramatic Arts Medical Clowning Program is the first academic and research program of its kind in the country, offering a groundbreaking opportunity to develop a new model for patient healing and wellness. While research studies have proven its effectiveness internationally, USC hopes to become a leading player by applying, proving, and advocating for the transformational impact of clowning in healthcare. Medical Clowns, Zachary Steel and Caitlyn Conlin, have both been clowning at LAC + USC County Hospital for the past two years. The practice, as perceived by the clown practitioners, staff and family members, has been extremely effective in lowering anxiety, reframing the hospitalization experience, and as a distraction tool. We are hoping to elevate the practice as a vital paramedical profession by proving the efficacy of the practice in this specific setting.

Internationally, the practice of medical clowning has becoming increasingly prevalent in hospital and community settings. The efficacy of the practice continues to be proven, all without undue risk to human subjects, when applied to a large spectrum of populations and settings. At Carmel Medical Center in Haifa, Israel, a study on the effect of medical clowning on reducing pain, crying, and anxiety in children aged 2 to 10 years old undergoing venous blood drawing proved the clowns were effective, safe, and had less negative effect on future blood draw examinations compared with control or use of topical anesthetic. Furthermore, integration of medical clowns in physical examination was shown to improve the overall experience of the child and the caregivers and help the pediatrician to perform a complete physical examination, with shorter duration of discomfort (0.2 +/- 0.6 minutes vs 1.6 +/- 2.0 minutes, p = 0.001); in the medical clown group, 94% of pediatricians reported that the medical clown improved their ability to perform a complete physical examination. Clowning has also successfully been used as a psychological distress buffer during anogenital examinations of sexually abused children.

While the international community has successfully studied the efficacy of the practice, the practice of medical clowning varies from country to country as the patient's response to different forms of humor and play varies. Culturally, clowns play a different role in the United States than they do elsewhere due to coulrophobia (fear of clowns) that has surfaced in the U.S. due to blockbuster movies. In 2017, an Israeli group published a study that showed that only 1.2% of hospitalized children were afraid of clowns. In contrast, according to a poll conducted by Morning Consult 42% of Americans said they were, in some capacity, afraid of clowns.

Participants will be randomized to either receive medical clowning intervention or no intervention. The total length of subject participation is the participant's one visit to the blood draw clinic.

Each participant randomized to the medical clowning arm will undergo one medical clowning session which consists of two medical clowns accompanying them before, during, and after venipuncture. The data collection procedures (surveys, recordings), are not experimental but will be performed exclusively for research purposes. Initial pre-intervention surveys will be administered in the waiting room to the participant and legal guardians before the blood draw procedure. Post-intervention surveys will be administered once the participant leaves the blood draw room. For both the intervention and non-intervention group, the nurses will communicate to the research assistant if the papoose was used. For both the intervention and non-intervention group, audio will begin recording the moment the participant steps into the blood draw room to later assess duration of crying. The detailed design of the study is as follows:

SCREENING & CONSENT FORM PHASE (15-20 minutes): Participants will be screened for eligibility based on the inclusion and exclusion criteria. After identifying eligible candidates, immediately following patient check-in at the clinic's front desk, the participant patient and legal guardian will receive a written overview of the study and will have time to ask questions regarding the purpose of the study and what's to be expected of them. If they agree to participate, participants aged 7-11 will be asked to give assent and all legal guardians will be asked to sign an Informed Consent Form. The participant and guardian will be given trial specific information. All referring physicians and nurses will be informed of their participants' enrollment. In the case that the participant and legal guardian are more proficient in Spanish than English, all of these forms and documents will be provided to them in Spanish.

PRE-INTERVENTION PHASE (WAITING ROOM) (15-20 minutes): All documents will be copied and distributed / filed, including copies to the family. The participant will be registered and randomized as per protocol. Initial pre-intervention surveys will be administered.

CLOWN INTRODUCTION PHASE (3-5 minutes): Participants and caregivers sit in a hallway before they are admitted into a blood draw room. For the intervention patient, once the survey is completed, the clowns will introduce themselves to the subjects and form an introductory bond. The clown will accompany the child to the blood draw room. For the non-intervention participant, no clown will be introduced and they will wait for the nurse to lead them into the blood draw room to continue usual care.

CLINICAL PHASE (variable duration, estimated 30-40 minutes, depending on routine medical care duration): For the intervention group, the nurse administers usual standard nursing care (vitals: blood pressure cuff, temperature reading, oxygen saturation, etc.). The clowns will work in complement, finding opportunities to connect and find play opportunities with the patient and caretakers to ease anxiety, lessen crying duration, and improve the overall experience. The clown engages with the participant and all caregivers in the room and attempts to divert their focus away from pain and reduce their anxiety levels through play, laughter, and imagination during venipuncture and other nursing care. Following the collection of blood samples by the nurses, the clowns will stay in the room to soothe and play a transitional role prior to returning to routine care with subsequent providers (e.g. doctor, social worker, dietician). For the non-intervention group, no clown will be present and the nurses will proceed with routine tests and blood draw. The nurse will use the papoose only if determined necessary to subdue the child during venipuncture. For both the intervention and non-intervention-groups, the nurses will communicate to the research assistant if the papoose was used. For both the intervention and non-intervention groups, audio will begin recording the moment a child steps into the blood draw room to later assess duration of crying.

POST-SURVEY PHASE (10-15 minutes): Post-intervention surveys will be administered.

MEDICAL STAFF FOLLOW UP PHASE: At the end of the entire study, the medical staff will be asked to answer a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Children whose treatment includes blood tests in the outpatient blood draw facility at LAC + USC Medical Center.

Exclusion Criteria:

* Participants will be excluded if they have severe developmental disabilities or are both blind and deaf.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
2-Item anxiety intensity measure | 30 minutes
  Compare the difference in self reported scores on the Children's Anxiety and Pain Scale 0-4 prior to and 0-4 following intervention, between control and experimental groups

SECONDARY OUTCOMES:
2-item pain intensity measure | 30 minutes
  Compare the difference in self reported scores on the Wong-Baker FACES Pain Rating Scale 0-4 prior to and 0-4 following intervention, between control and experimental groups

CONTACTS AND LOCATIONS:
Overall Officials: Brent Blair, Principal Investigator — University of Southern California
Locations (1):
- LAC+USC Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedler S, Glasser S, Azani L, Freedman LS, Raziel A, Strassburger D, Ron-El R, Lerner-Geva L. The effect of medical clowning on pregnancy rates after in vitro fertilization and embryo transfer. Fertil Steril. 2011 May;95(6):2127-30. doi: 10.1016/j.fertnstert.2010.12.016. Epub 2011 Jan 6. PMID 21211796
- [Background] Dafna Tener, Nessia Lang-Franco, Shoshi Ofir & Rachel Lev-Wiesel (2012) The Use of Medical Clowns as a Psychological Distress Buffer During Anogenital Examination of Sexually Abused Children, Journal of Loss and Trauma, 17:1, 12-22, DOI: 10.1080/15325024.2011.578025
- [Background] Meiri N, Ankri A, Hamad-Saied M, Konopnicki M, Pillar G. The effect of medical clowning on reducing pain, crying, and anxiety in children aged 2-10 years old undergoing venous blood drawing--a randomized controlled study. Eur J Pediatr. 2016 Mar;175(3):373-9. doi: 10.1007/s00431-015-2652-z. Epub 2015 Oct 16. PMID 26475347
- [Background] Meiri N, Ankri A, Ziadan F, Nahmias I, Konopnicki M, Schnapp Z, Itzhak Sagi O, Hamad Saied M, Pillar G. Assistance of Medical Clowns Improves the Physical Examinations of Children Aged 2-6 Years. Isr Med Assoc J. 2017 Dec;19(12):786-791. PMID 29235739
- [Background] Goldberg A, Stauber T, Peleg O, Hanuka P, Eshayek L, Confino-Cohen R. Medical clowns ease anxiety and pain perceived by children undergoing allergy prick skin tests. Allergy. 2014 Oct;69(10):1372-9. doi: 10.1111/all.12463. Epub 2014 Aug 4. PMID 24943088
- [Background] Rimon A, Shalom S, Wolyniez I, Gruber A, Schachter-Davidov A, Glatstein M. Medical Clowns and Cortisol levels in Children Undergoing Venipuncture in the Emergency Department: A Pilot Study. Isr Med Assoc J. 2016 Nov;18(11):680-683. PMID 28466619